CLINICAL TRIAL: NCT02324270
Title: Randomized, Double-Blind, Multiple-Center, Placebo-Controlled Study Comparing the Safety and Efficacy of Generic Diclofenac Epolamine to Flector® Patch in the Treatment of Acute Pain Due to Minor Ankle Sprain
Brief Title: Safety and Efficacy of Generic Diclofenac Epolamine Acute Pain Due to Minor Ankle Sprain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DICLO-13-01
Record Dates: First submitted 2014-12-08; First posted 2014-12-24 (Estimated); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Ankle Sprain
Keywords: Pain due to ankle sprain
MeSH Terms: conditions — Ankle Injuries | interventions — diclofenac hydroxyethylpyrrolidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diclofenac epolamine (Active Comparator): Flector® (Diclofenac Epolamine Topical Patch 1.3%) (Pfizer)
  Interventions: Drug: Diclofenac epolamine
- generic diclofenac epolamine patch (Experimental): Generic Diclofenac Epolamine Topical Patch 1.3% (Watson Laboratories, Inc.)
  Interventions: Drug: Diclofenac epolamine
- Placebo (Placebo Comparator): Placebo patch of the test product (Watson Laboratories, Inc.); Identical in appearance and formulated as the test product, omitting the active ingredient, diclofenac epolamine
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Diclofenac epolamine — Diclofenac epolamine in a topical patch formulation; applied to the area of sprained ankle; to treat pain associated with a mild ankle sprain
  Other Names: Flector Patch
  Arms: Diclofenac epolamine; generic diclofenac epolamine patch
Other: Placebo — Topical patch not containing diclofenac epolamine applied to the area of sprained ankle; to treat pain associated with a mild ankle sprain
  Other Names: Vehicle control
  Arms: Placebo

SUMMARY:
To demonstrate the therapeutic efficacy of a generic diclofenac epolamine patch against Flector patch in the treatment of pain in subjects with minor ankle sprain

DETAILED DESCRIPTION:
To evaluate the therapeutic equivalence and safety of generic diclofenac epolamine 1.3% patch (Watson Laboratories, Inc.) and Flector® (diclofenac epolamine 1.3% patch) (Pfizer) in the treatment of acute pain due to minor ankle sprain.

To demonstrate the superiority of the efficacy of the test and reference products over that of the vehicle control in the treatment of acute pain due to minor ankle sprain.

To access application site reactions and patch adhesion between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Non pregnant females, 18-65 years of age
2. Signed informed consent obtained that meets all criteria of current FDA and Health Insurance Portability and Accountability Act regulations
3. Subject has a diagnosis of uncomplicated acute minor ankle sprain: Grade I and II (as defined by the America Academy of Orthopedic Surgeons AAOS)
4. Ankle sprain must have occurred < 48 hours before study entry with baseline pain score of > 50 mm on a 100 mm Visual Analog Scale (VAS) upon active mobilization
5. Female subjects of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 1 year), in addition to having a negative urine pregnancy test, must be willing to use an acceptable form of birth control during the study from the day of the first dose administration to 30 days after the last administration of study drug. For the purpose of this study the following are considered acceptable methods of birth control: oral or injectable contraceptives, contraceptive patches, Depo-Provera® (on stable treatment for at least 3 months) NuvaRing® (vaginal contraceptive); Implanon™ (contraceptive implant) double barrier methods (e.g. condom and spermicide), intrauterine device, or abstinence with a 2nd acceptable method of birth control, should the patient become sexually active. A sterile sexual partner is NOT considered an adequate form of birth control.
6. All male subjects must agree to use accepted methods of birth control with their partners, from the day of the first dose administration to 30 days after the last administration of study drug. Abstinence is an acceptable method of birth control. Female partners should use an acceptable method of birth control as described in Item Number 5.
7. Subject is free from any systemic or dermatologic disorder that, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events.
8. Subject shows willingness and capability to cooperate to the extent and degree required by the protocol.
9. Subject is willing to refrain from using any other pain medication during their participation.

Exclusion Criteria:

1. Pregnant or breastfeeding female.
2. Sprain occurred > 48 hours prior to study enrollment.
3. Ankle sprain requires an orthopedic or surgical treatment.
4. Ankle sprain treated prior to study entry by topical, oral, or parenteral nonsteroidal antiinflammatory drug (NSAID), physiotherapy, ultrasound, physical therapy or acupuncture.
5. Baseline self-evaluation of pain on active mobilization by the VAS < 50 mm.
6. Non-intact or damaged skin within the area to be treated, e.g., eczema, psoriasis, exudative, dermatitis, infected lesion, burn or wound.
7. Medical history of asthma, urticaria, angioedema, bronchospasm, ulcer disease, gastrointestinal bleeding, hypertension, edema, heart failure or cardiovascular disease.
8. Medical history of any chronic pain disorder.
9. Coagulation defects.
10. Severe cardiac, renal or hepatic impairment.
11. Severe systemic disease (e.g., cancer, severe acute infection).
12. Use within one month prior to randomization of 1.) immunomodulators or immunosuppressive therapies, 2.) interferon, 3.) oral or parenteral corticosteroids or 4.) cytotoxic drugs.
13. Use within 7 days prior to randomization of any topical agents on the affected ankle.
14. Use within 7 days prior to randomization of topical, oral or parenteral treatment with NSAIDs or aspirin.
15. Use within 12 hours prior to randomization of an analgesic. Eg. Acetaminophen (Tylenol®).
16. Known allergy or hypersensitivity to diclofenac, aspirin or other NSAIDs, or any excipient in the test product or brand product (Flector).
17. History of uncontrolled chronic or acute concomitant disease which, in the Investigator's opinion, would contraindicate study participation or confound interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Lau, PhD, Study Director — Actavis Inc.
Locations (31):
- United States (31):
  - Site 21, Birmingham, Alabama
  - Site 24, Goodyear, Arizona
  - Site 08, Carlsbad, California
  - Site 05, Ventura, California
  - Site 16, Clinton, Connecticut
  - Site 03, Riverton, Connecticut
  - Site 11, Daytona Beach, Florida
  - Site 09, DeLand, Florida
  - Site 14, Miami, Florida
  - Site 07, Miami, Florida
  - Site 13, Miami, Florida
  - Site 02, West Palm Beach, Florida
  - Site 26, Lexington, Kentucky
  - Site 12, Gretna, Louisiana
  - Site 23, Kalamazoo, Michigan
  - Site 41, Traverse City, Michigan
  - Site 10, Omaha, Nebraska
  - Site 29, Berlin, New Jersey
  - Site 18, Brooklyn, New York
  - Site 19, Cincinnati, Ohio
  - Site 30, Columbus, Ohio
  - Site 35, Oklahoma City, Oklahoma
  - Site 37, Downingtown, Pennsylvania
  - Site 27, State College, Pennsylvania
  - Site 15, Austin, Texas
  - 04, El Paso, Texas
  - Site 34, Houston, Texas
  - Site 36, Lake Jackson, Texas
  - Site 22, San Antonio, Texas
  - Site 31, Danville, Virginia
  - Site 06, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The populations for this study included the Safety Population, the Per-Protocol Population (PP) and the modified Intent-to-treat (mITT) population.
Groups:
- Diclofenac Epolamine Patch (Test Product): Generic Diclofenac Epolamine Topical Patch 1.3% (Watson Laboratories, Inc.)
  Diclofenac epolamine: Diclofenac epolamine in a topical patch formulation; applied to the area of sprained ankle; to treat pain associated with a mild ankle sprain
- Flector (Reference Product): Flector® (Diclofenac Epolamine Topical Patch 1.3%) (Pfizer)
  Diclofenac epolamine: Diclofenac epolamine in a topical patch formulation; applied to the area of sprained ankle; to treat pain associated with a mild ankle sprain
Period: Overall Study
Arm/Group | Diclofenac Epolamine Patch (Test Product) | Flector (Reference Product) | Placebo
Started | 218 | 219 | 221
Safety Population | 214 | 216 | 217
mITT Population | 214 | 216 | 217
PP Population | 180 | 177 | 171
Completed | 213 | 212 | 216
Not Completed | 5 | 7 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 3 | 4
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Non Compliance with Study Drug | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Epolamine Patch (Test Product) | Flector (Reference Product) | Placebo | Total
Number analyzed (Participants) | 214 | 216 | 217 | 647
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (12.1) | 34.9 (12.5) | 35.5 (13.3) | 35.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 79 | 82 | 246
  Male | 129 | 137 | 135 | 401
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 86 | 78 | 83 | 247
  Not Hispanic or Latino | 128 | 138 | 134 | 400
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 5 | 11
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 60 | 59 | 71 | 190
  White | 147 | 149 | 140 | 436
  More than one race | 0 | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 214 | 216 | 217 | 647
Height (cm) [Mean (Standard Deviation); unit: cm] | 171.44 (10.74) | 173.28 (10.80) | 172.17 (9.72) | 172.30 (10.44)
Weight (kg) [Mean (Standard Deviation); unit: Kg] | 81.73 (19.86) | 83.34 (17.11) | 83.97 (20.10) | 83.02 (19.07)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) Scores at Baseline and Post Treatment
Description: To evaluate the therapeutic equivalence (90% CI) of generic diclofenac epolamine 1.3% patch (Watson Laboratories, Inc.) and Flector® (diclofenac epolamine 1.3% patch) (Pfizer) using a 100mm VAS scoring in the treatment of acute pain due to minor ankle sprain (in the per protocol population); changes from baseline.
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as lower values of 'no pain at all' and higher values relating to 'pain as bad as it could be' .
  Percent improvement in VAS score is the percentage part of - change from baseline in VAS / Baseline VAS.
Time Frame: Baseline, 3 days
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diclofenac Epolamine Patch (Test Product) | Flector (Reference Product)
Number analyzed (Participants) | 180 | 177
score on a scale
  Baseline | 68.56 (11.03) | 69.03 (10.90)
  72 Hours after Initial treatment | 25.34 (17.35) | 25.78 (18.50)
  Change from Baseline | -43.22 (18.94) | -43.25 (20.71)
Statistical Analysis 1: Comparison: Diclofenac Epolamine Patch (Test Product) vs Flector (Reference Product); Test type: Equivalence — If the 90% CI for the ratio of mean changes between test and reference products was contained within the interval, [0.80,1.25], then the products were considered to be equivalent; Ratio = 1.01, 90% CI 2-sided [0.94 to 1.08]

2. Secondary Outcome: Visual Analogue Scale (VAS) Scores at Baseline and Post Treatment
Description: To demonstrate the superiority (P<0.05) of the efficacy of the test and reference products over that of the vehicle control in the treatment of acute pain utilizing a 100 mm VAS (in the mITT population) - changes from baseline.
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as lower values of 'no pain at all' and higher values relating to 'pain as bad as it could be' .
Time Frame: Baseline, 3 days
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diclofenac Epolamine Patch (Test Product) | Flector (Reference Product) | Placebo
Number analyzed (Participants) | 214 | 216 | 217
score on a scale
  Baseline | 68.75 (11.27) | 68.93 (10.94) | 70.09 (11.37)
  72 hours after Initial treatment | 25.83 (18.19) | 26.16 (18.47) | 27.16 (18.18)
  Change from baseline | -42.91 (19.04) | -42.80 (20.73) | -42.88 (21.66)
Statistical Analysis 1: Comparison: Diclofenac Epolamine Patch (Test Product) vs Placebo; Test type: Superiority; p = 0.01, ANCOVA
Statistical Analysis 2: Comparison: Flector (Reference Product) vs Placebo; Test type: Superiority; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline up to 3 days (72 hours)
Description: Adverse events were collected from participants who were randomized and received at least one dose of study drug
Arm/Group | Diclofenac Epolamine Patch (Test Product) | Flector (Reference Product) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/214 | 0/216 | 0/217
Serious Adverse Events (participants affected / at risk) | 0/214 | 0/216 | 0/217
Other Adverse Events (participants affected / at risk) | 17/214 | 20/216 | 22/217
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac Epolamine Patch (Test Product) (N=214) | Flector (Reference Product) (N=216) | Placebo (N=217)
Headache (Nervous system disorders) | 3 | 1 | 6
Dizziness (Nervous system disorders) | 1 | 2 | 1
Paraesthesia (Nervous system disorders) | 2 | 1 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 1
Application site pruritus (General disorders) | 1 | 4 | 5
Pain (General disorders) | 0 | 1 | 2
Application site pain (General disorders) | 0 | 0 | 2
Swelling (General disorders) | 0 | 1 | 1
Application site burn (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory fatigue (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 2 | 0
Heart rate increased (Investigations) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.